CLINICAL TRIAL: NCT06154148
Title: Comparison of Two Different Skin-to-skin Contact Techniques: Sustained Diagonal Flexion (SDF) With Sling Versus Traditional Prone Position With Headband During Skin-to-skin Care Session
Brief Title: Comparison of Two Different Skin-to-skin Contact Techniques: Sustained Diagonal Flexion vs. Traditional
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Dorottya kelen, Head of Neonatal Unit, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P2021/338 B4062021000175
Record Dates: First submitted 2021-09-13; First posted 2023-12-01 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Skin-to-skin; Preterm Birth
Keywords: Kangaroo Care; Skin-to-skin; Sustained diagonal flexion; skin-to-skin contact time; Joint mobility and muscular tension assessment; Preterm; Family centered care
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sustained Diagonal Flexion positioning (Experimental): This position is a semi reclined positioning, the premature infant is off-center and semi-reclined on the mother's chest its body-axis is slightly flexed, with the limbs retracted in a preventive posture and the head in line with the body axis, moderately externally rotated hips in flexion-abduction, with adducted shoulders. The infants's head turns toward the mother's face and is located between the nipple and the clavicle. Their arms and legs are flexed, in a naturally adopted asymmetrical tonic neck posture, according to the infants's term and comfort. The infant is naked and positioned inside the mother's clothes.
  Interventions: Procedure: Sustained Diagonal Flexion positioning
- Traditional prone position (Active Comparator): The infants are placed vertically between the mother's breasts firmly attached to the chest and below their clothes.
  Interventions: Procedure: Traditional prone position

INTERVENTIONS:
Procedure: Sustained Diagonal Flexion positioning — This position is a semi reclined positioning, the infant is off-center and semi-reclined on the mother's chest its body-axis is slightly flexed, with the limbs retracted in a preventive posture and the head in line with the body axis, moderately externally rotated hips in flexion-abduction, with adducted shoulders. The infant's head turns toward the mother's face and is located between the nipple and the clavicule. Their arms and legs are flexed,in a naturally adopted asymmetrical tonic neck posture, according to the infant's term and comfort. The infant is naked and positioned inside the mother's clothes.
  Other Names: FDS
  Arms: Sustained Diagonal Flexion positioning
Procedure: Traditional prone position — The infant is placed vertically between the mother's breasts firmly attached to the chest and below their clothes.
  Arms: Traditional prone position

SUMMARY:
This is a prospective, controlled randomized study designed to compare the effects of two methods of skin-to-skin positioning of preterm infants: the prone positioning method currently used (according to the World Health Organization's recommendations) and the recent "sustained diagonal flexion" method (SDF) on the daily duration of skin-to-skin contact.

DETAILED DESCRIPTION:
This is a prospective, controlled, randomized, non-blinded trial, recruiting premature infants between 27- 34 weeks of gestational age during the first 4 days of life.

80 parent-infant dyads will be recruited in the Department of Neonatology (GA between 27 and 34 weeks) and randomly divided in two groups. Each dyads will be assigned to one of the two skin-to-skin positions.

The study aims to investigate if the sustained diagonal flexion method (SDF) provides additional benefits for both the child and their parents, such as increase in daily skin-to-skin time and its continuation after discharge.

The investigators will analyze the daily duration of skin-to-skin, the cardiorespiratory stability of the child (number of incidents recorded by standard monitoring), the presence of pain during: installation /skin-to-skin/ after the return to the incubator, the continuation of skin-to-skin, breastfeeding after discharge, the risk of postpartum depression in the mother, parental stress, joint mobility and muscle tension of the child and their parents, and also the comfort and satisfaction with the type of skin-to-skin.

ELIGIBILITY:
Inclusion Criteria:

* Premature infant born between 27 and 34 weeks of gestational age
* Aged between 24 hours and maximum 4 days at the beginning of the study
* Approval from the neonatologist in charge of the patient to participate in the study
* Informed consent of the parents to participate in the study
* At least one of the two parents must have a good knowledge of French.

Exclusion Criteria:

* Infant with severe secondary neurological or medical conditions, e.g., neurological deficits due to vascular hemorrhage (grade III or IV)
* Infant or parent who requires or has required surgery during their neonatal stay
* Triplets
* Parent who suffers from a physical disability or severe psychological illness, a psychosocial situation that does not allow skin-to-skin care
* Infant with an arterial line

Ages: 24 Hours to 4 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Daily duration of skin-to-skin during postnatal hospitalisation | during hospitalisation
  Investigate the effect of skin-to-skin position of premature infants in supported diagonal flexion (SDF) by a sling on daily duration of skin to skin contact during hospitalization (Measured in minutes per day. )
Continuation of skin-to-skin after discharge | 6 months
  Time spent in a sling by 6 months of age. (Measured in minutes per day)

SECONDARY OUTCOMES:
Breastfeeding at discharge and at 1, 3, 6 month of age | 6 months
  Breastfeeding at discharge and duration of breastfeeding after discharge; Continuation of breastfeeding (exclusive or mixed), use of breast pump and reasons for stopping breastfeeding (work - other) will be collected by telephone interview from parents at 1, 3 and 6 months after discharge.
Cardiovascular stability of the infant | 3-12 weeks
  Occurrence of apnea, bradycardia, and desaturation episodes; Number of incidents will be recorded from the monitoring at installation, during the skin-to-skin time and during the de-installation (number of bradycardias, apneas, desaturations, hypothermia < 36°C). Any comments from the caregiver or parent will also be noted. (Measured in episodes/hour)
Physiological parameters via Stability of the Cardiorespiratory System in Premature Infants (SCRIP) score | 3-22 days
  Between day 3 - 7 of life, day 10 - 12 of life and day 18-22 of life a specific recording of the physiological parameters via the Stability of the Cardiorespiratory System in Premature Infants (SCRIP) score will be carried out two hours before, during the first two hours, and two hours after the end of the intervention. The SCRIP score measure three parameters of the cardiorespiratory stability of the infants. (Score between 0-6, low score indicates instability, high score indicates stability.
Physiological parameters via Newborn Infant Parasympathetic Evaluation (NIPE) scores | 3-22 days
  Between day 3 - 7 of life, day 10 - 12 of life and day 18-22 of life the NIPE (Newborn Infant Parasympathetic Evaluation) monitoring will be installed, the values taken will be those given 30 minutes before the skin-to-skin, the first hour of the skin-to-skin and 30 minutes after the skin-to-skin. The NIPE monitor provides an objective pain 'index' from 0 to 100. Lower indices reflect more pain, whereas higher indices indicate less pain.
Comfort-Behavior pain scale (Comfort-B) score measuring pain and comfort of the premature infant before during and after skin-to-skin contact | 3-12 days
  The "Comfort-Behavior" pain scale will be used 10 minutes after the installation. Immediately after the end of the session, parents will be given a satisfaction scale regarding the positioning experience and comfort, as well as a body chart on which the parent can note the areas where he or she experienced pain during the session. The Comfort-B score values for 6 items are scored between 1 and 5, generating scores between 6 and 30 points. Scores between 6 and 10 indicate oversedation; scores between 11 and 23 indicate a moderately sedated patient; and scores between 24 and 30 indicate little sedation.
Premature Infant Pain Profile-Revised (PIPP-R) pain score measuring pain and comfort of the premature infant before during and after skin-to-skin contact | 3-12 days
  Between day 3 - 7 of life, and day 10 - 12 of life the Premature Infant Pain Profile-Revised (PIPP-R) pain scale will be performed when the child is put in the sling (or headband). PIPP-R is scored for 7 items on a 4-point scale (0, 1, 2, 3) , and are summed for a total pain intensity score between 6 and 28, higher score indicates more pain.
Position of joints and muscle tone observed by osteopath or physiotherapist and evaluated by joint, posture and muscle tone assessment -JPMA established by the investigators | 2 days-12 weeks
  -Between day 2-6 of life and at hospital discharge, an osteopath or a physiotherapist, blind to the assignment of groups, will carry out a global observation of the child's posture, joint mobility and muscular tension assessment (JPMA), according to a questionnaire - predefined scale established by the investigators (Appendix IV). This assessment will be performed gently, when the baby is awake in the presence of the nurse in charge of the infant as well as the infant's parents if they so wish. This newly developed assessment scale is based upon existing scales developed for elder infants. Between day 18-22 of life, JPMA will be performed again by a physiotherapist or osteopath. At the same time, an evaluation of the physiological parameters during the skin-to-skin by means of the SCRIP score will be performed. At discharge, the JPMA will be performed too. Score is between 0-4, 4 being the worst
Parental psychological wellbeing - French version of the Parental Stressor Scale (PSS) | 1 day-22 days
  Immediately after signing the consent form, and at day 18-22 of admission, the French version of the Parental Stressor Scale (PSS) will be given to each parent to complete individually. Each envelope containing the questionnaires will then be sealed by the parent and given to the examiners. The envelope will only be opened at the end of the child's care and only for the purpose of collecting data for the study. Before discharge, parents will be asked to complete PSS again as well as the visual analog scale regarding satisfaction and interactions with their infant during skin-to-skin contact. Score between 0-40, high score indicate worsening stress.
Parental psychological wellbeing - the Edinburgh Postnatal Depression Scale (EPDS) | 1 day-22 days
  Immediately after signing the consent form, and at day 18-22 of admission, the Edinburgh Postnatal Depression Scale (EPDS) will be given to each parent to complete individually. Each envelope containing the questionnaires will then be sealed by the parent and given to the examiners. The envelope will only be opened at the end of the child's care and only for the purpose of collecting data for the study. Before discharge, parents will be asked to complete EPDS again as well as the visual analog scale regarding satisfaction and interactions with their infant during skin-to-skin contact. Score between 0-30, 7-13 mild, 14-19 moderate 20-30 severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Dorottya Kelen, Principal Investigator — Head of Neonatal Unit
Locations (1):
- Neonatal Unit Hopital Erasme, Brussels, Anderlecht, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] WHO Recommendations on Interventions to Improve Preterm Birth Outcomes. Geneva: World Health Organization; 2015. Available from http://www.ncbi.nlm.nih.gov/books/NBK321160/ PMID 26447264
- [Result] Conde-Agudelo A, Diaz-Rossello JL. Kangaroo mother care to reduce morbidity and mortality in low birthweight infants. Cochrane Database Syst Rev. 2016 Aug 23;2016(8):CD002771. doi: 10.1002/14651858.CD002771.pub4. PMID 27552521
- [Result] Puthussery S, Chutiyami M, Tseng PC, Kilby L, Kapadia J. Effectiveness of early intervention programs for parents of preterm infants: a meta-review of systematic reviews. BMC Pediatr. 2018 Jul 9;18(1):223. doi: 10.1186/s12887-018-1205-9. PMID 29986683
- [Result] Coskun D, Gunay U. The Effects of Kangaroo Care Applied by Turkish Mothers who Have Premature Babies and Cannot Breastfeed on Their Stress Levels and Amount of Milk Production. J Pediatr Nurs. 2020 Jan-Feb;50:e26-e32. doi: 10.1016/j.pedn.2019.09.028. Epub 2019 Oct 28. PMID 31672261
- [Result] Pados BF, Hess F. Systematic Review of the Effects of Skin-to-Skin Care on Short-Term Physiologic Stress Outcomes in Preterm Infants in the Neonatal Intensive Care Unit. Adv Neonatal Care. 2020 Feb;20(1):48-58. doi: 10.1097/ANC.0000000000000596. PMID 30893092
- [Result] Buil A, Carchon I, Apter G, Laborne FX, Granier M, Devouche E. Kangaroo supported diagonal flexion positioning: New insights into skin-to-skin contact for communication between mothers and very preterm infants. Arch Pediatr. 2016 Sep;23(9):913-20. doi: 10.1016/j.arcped.2016.04.023. Epub 2016 Jul 4. PMID 27388909
- [Result] Vaivre-Douret L, Ennouri K, Jrad I, Garrec C, Papiernik E. Effect of positioning on the incidence of abnormalities of muscle tone in low-risk, preterm infants. Eur J Paediatr Neurol. 2004;8(1):21-34. doi: 10.1016/j.ejpn.2003.10.001. PMID 15023372
- [Result] Ferrari F, Bertoncelli N, Gallo C, Roversi MF, Guerra MP, Ranzi A, Hadders-Algra M. Posture and movement in healthy preterm infants in supine position in and outside the nest. Arch Dis Child Fetal Neonatal Ed. 2007 Sep;92(5):F386-90. doi: 10.1136/adc.2006.101154. Epub 2007 Mar 7. PMID 17344252
- [Result] Stevens BJ, Gibbins S, Yamada J, Dionne K, Lee G, Johnston C, Taddio A. The premature infant pain profile-revised (PIPP-R): initial validation and feasibility. Clin J Pain. 2014 Mar;30(3):238-43. doi: 10.1097/AJP.0b013e3182906aed. PMID 24503979